CLINICAL TRIAL: NCT05068557
Title: Dietary Intervention Supplemented With PUFA Omega-3 Fatty Acids on the Pro-resolving Capacity in Subjects With Obesity.
Brief Title: EPICO: (Study for the Pro-resolution of Chronic Inflammation in Obesity. Original Acronym From Spanish)
Acronym: EPICO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Guadalajara (Other)
Responsible Party: Principal Investigator, ERIKA MARTINEZ-LOPEZ, PhD, University of Guadalajara
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CI03221
Record Dates: First submitted 2021-09-22; First posted 2021-10-06 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-10

CONDITIONS: Obesity; Chronic Inflammation
Keywords: PUFA omega 3; Obesity; Low-grade chronic inflammation; Specialized-proresolving mediators; Inflammation resolution
MeSH Terms: conditions — Obesity | interventions — Fish Oils

STUDY DESIGN:
Intervention Model Description: Double-blind randomized parallel clinical trial
Who Masked: Participant, Investigator
Masking Description: Both type of capsules were deposited in equally labeled flaks under sterile conditions. Every flask was identified and tagged with a specific number by an associate researcher who is not involved in the recruitment, attention, or follow-up of the enrolled subjects. Finally, block randomization was the selected technique for this purpose.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): Dietary plan with a mild calorie restriction and adjusted in PUFA omega-3/omega-6 ratio (4:1) along with fish oil (3 capsules daily. Containing EPA+DHA: 1.8 g). (n=40)
  Interventions: Dietary Supplement: Dietary plan along with fish oil capsules (3 capsules daily. Containing EPA+DHA: 1.8 g).
- Control group (Placebo Comparator): Dietary plan with a mild calorie restriction and adjusted in PUFA omega-3/omega-6 ratio (4:1) along with chia/linseed oil (3 capsules daily. Containing ALA 1.6 g). (n=40)
  Interventions: Dietary Supplement: Dietary plan along with chia/linseed oil capsules (3 capsules daily. Containing ALA 1.6 g).

INTERVENTIONS:
Dietary Supplement: Dietary plan along with fish oil capsules (3 capsules daily. Containing EPA+DHA: 1.8 g). — Subects within the Intervention group will be provided with a dietary plan along with fish oil capsules. Subjects will be asked to consume three capsules per day. Every capsule contains: EPA+DHA: 1.8 g.
  Other Names: Dietary intervention along with fish oil
  Arms: Intervention group
Dietary Supplement: Dietary plan along with chia/linseed oil capsules (3 capsules daily. Containing ALA 1.6 g). — Subects within the Intervention group will be provided with a dietary plan along with fish oil capsules. Subjects will be asked to consume three capsules per day. Every capsule contains: ALA 1.6 g).
  Other Names: Placebo
  Arms: Control group

SUMMARY:
Omega-3 fatty acids, especially EPA and DHA have long been acknowledged for their capacity to counteract inflammatory responses in the human body. Understanding the impact of the dietary intake of these fatty acids along with others (such as ARA) involved in inflammation is essential for prevention and treatment of chronic non-communicable diseases as it is obesity and its comorbidities.

The role that the EPA and DHA play in the inflammatory processes can be understood by studying the capacity of certain immune cells and their genetic background to respond under the constant exposure to an adjusted diet in omega-6/omega-3 fatty acids in individuals with obesity.

DETAILED DESCRIPTION:
A total of 80 subjetcs will be invited to be enrolled in a nutrigenomics/nutrigenetics study approaching the properties of a dietary plan (mild calorie restriction and adjusted at an omega-6/omega-3 fatty acids ratio of 4:1, and supplemented with fish oil rich in EPA and DHA or placebo).

This double blind, randomized, parallel clinical trial will consist in a 12-week intervention with recurrent visits every 4 weeks. Subjects will be required to follow the dietary plan provided in a recipee book produced and edited by our research group along with a capsule in every major meal (breakfast, lunch, and dinner) for 12 weeks. In every visit, all subects will undergo a body composition analysis as well as blood tests that include: total cell count, glucose and lipid homeostasis, serum inflammatory markers, DNA extraction for genetic tests (SNPs involved in inflammation), isolation and ex vivo stimulation of neutrophils, determination of and isolation of PBMCs for further analysis of gene expression and protein abundance.

This study proposes three distinct but closely related approaches for reaching a further understanding of the actions of EPA and DHA intake:

1. Through the conversion of EPA and DHA to specialized pro-resolving mediators (SPMs) such as resolvins (E and D) determined by an ex vivo assay
2. Through the study of the involved enzyme coding-genes in the previously mentioned conversion
3. Through the study of the activation of specific membrane receptors (FFAR4)

All these approaches will have in common the correlation with serum inflammatory markers (TNF alpha, MCP1, IL-6, and IL-10).

Once the project is finished, the research strategies for new studies will be improved. In the same way, the application of the knowledge generated in it will be encouraged towards the health care of patients with obesity who could attend our service on future occasions. Finally, we would disseminate the knowledge generated in our institutional community, which would increase the impact of the project.

In summary, the impact is divided into the following points:

* Identification of genetic markers relevant to the treatment of obesity and its comorbidities
* Bases for new strategies aimed at reducing chronic low-grade inflammation inherent in obesity
* Useful information on gene-nutrient interaction for the public and private sector in the field of genetic testing
* Study population benefited from the results of the intervention and the information of their genetic and biochemical profiles Data from this study would strengthen the inflammatory knowledge of obesity comorbidities from distinct standpoints

ELIGIBILITY:
Inclusion Criteria:

* 25-59 years of age, both sexes
* Subjects who agree to participate in the study and all signed informed consent
* BMI 30 kg/m2 - 39.9 kg/m2
* Waist circumference >88 cm for females; >102 cm for males

Exclusion Criteria:

* Currently consuming any of the following drugs: NSAIDS, anticoagulants, hypoglycemic, oR hypolipemic drugs
* Diagnosed autoimmune diseases
* Diagnosed cancer
* Pregnancy and breastfeeding
* Allergy to chia, linseed or fish oil
* Subjects who wish to abandon the study

Ages: 25 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-09-24 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Resolvin E1 and D1 secretion under stimulation conditions (ex vivo). | 12 weeks
  Stimulation of neutrophils from subjects who underwent a dietary plan (mild calorie restriction along with an omega-6/omega-3 adjusted ratio and supplemented with fish oil or placebo) and their correlation with inflammatory markers (serum TNF alpha, IL-6, MCP1, and IL-10). The major markers of change are resolvin E1 and resolvin D1 (RvE1 and RvD1).
Genetic analysis of Single Nucleotide Polymorphism (SNPs) involved in the synthesis of specialized pro-resolving mediators (SPMs). | 12 weeks
  Subjects who underwent a dietary plan (mild calorie restriction along with an omega-6/omega-3 fatty acids adjusted ratio and supplemented with fish oil or placebo) will be genotyped based on inflammatory genetic variants: CYP4F3 (rs1805042), PTGS2 (rs5275, rs20417, and rs689466) y ALOX15 (rs11568131) and their correlation with the (ex vivo) secretion of Resolvin E1 and D1 and with inflammatory markers (serum TNF alpha, IL-6, MCP1, and IL-10).
Analysis of the activation of FFAR4 in PBMCs | 12 weeks
  Analysis through immunoprecipitation and immunoblotting to determine the activation of FFAR4 in PBMCs and their correlation with inflammatory markers (serum TNF alpha, IL-6, MCP1, and IL-10). Subjects who underwent a dietary plan (mild calorie restriction along with an omega-6/omega-3 fatty acids adjusted ratio and supplemented with fish oil or placebo)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Guadalajara (CUCS), Guadalajara, Jalisco, Mexico

REFERENCES:
- [Background] Rasic-Milutinovic Z, Perunicic G, Pljesa S, Gluvic Z, Sobajic S, Djuric I, Ristic D. Effects of N-3 PUFAs supplementation on insulin resistance and inflammatory biomarkers in hemodialysis patients. Ren Fail. 2007;29(3):321-9. doi: 10.1080/08860220601184092. PMID 17497447
- [Background] Polus A, Zapala B, Razny U, Gielicz A, Kiec-Wilk B, Malczewska-Malec M, Sanak M, Childs CE, Calder PC, Dembinska-Kiec A. Omega-3 fatty acid supplementation influences the whole blood transcriptome in women with obesity, associated with pro-resolving lipid mediator production. Biochim Biophys Acta. 2016 Nov;1861(11):1746-1755. doi: 10.1016/j.bbalip.2016.08.005. Epub 2016 Aug 12. PMID 27531277
- [Background] Souza PR, Marques RM, Gomez EA, Colas RA, De Matteis R, Zak A, Patel M, Collier DJ, Dalli J. Enriched Marine Oil Supplements Increase Peripheral Blood Specialized Pro-Resolving Mediators Concentrations and Reprogram Host Immune Responses: A Randomized Double-Blind Placebo-Controlled Study. Circ Res. 2020 Jan 3;126(1):75-90. doi: 10.1161/CIRCRESAHA.119.315506. Epub 2019 Dec 12. PMID 31829100
- [Background] Barden A, Shinde S, Tsai IJ, Croft KD, Beilin LJ, Puddey IB, Mori TA. Effect of weight loss on neutrophil resolvins in the metabolic syndrome. Prostaglandins Leukot Essent Fatty Acids. 2019 Sep;148:25-29. doi: 10.1016/j.plefa.2019.07.001. Epub 2019 Jul 3. PMID 31492430